CLINICAL TRIAL: NCT01357174
Title: Protocol for ROTATEQ™ Post-Marketing Surveillance
Brief Title: ROTATEQ™ Post-Marketing Surveillance in the Philippines
Status: Terminated | Type: Observational
Why Stopped: Merck Sharp & Dohme Corp (MSD) received exemption from PFDA on conduct of post-marketing surveillance (PMS) study
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: V260-046
Record Dates: First submitted 2011-05-18; First posted 2011-05-20 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Rotavirus Infections; Gastroenteritis
MeSH Terms: conditions — Rotavirus Infections; Gastroenteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Participants: Infants who were vaccinated with ROTATEQ™

SUMMARY:
This study will collect demographic and safety information on the use of ROTATEQ™ in the Philippines.

ELIGIBILITY:
Inclusion Criteria:

* Received ROTATEQ™

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants in the Philippines who received ROTATEQ.™ Information will be provided by the physicians who administered the vaccine.
Sampling Method: Non-Probability Sample
Enrollment: 915 (Actual)
Dates: Start 2007-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events following administration of ROTATEQ™ | Three-year period following vaccine marketing approval (August 2007 to August 2010)